CLINICAL TRIAL: NCT00000790
Title: Thalidomide for Treatment of Oral and Esophageal Aphthous Ulcers and HIV Viremia in Patients With HIV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Andrulis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 251; 11228 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Stomatitis, Aphthous
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Thalidomide; Stomatitis, Aphthous
MeSH Terms: conditions — HIV Infections; Stomatitis, Aphthous; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
PRIMARY: To evaluate the effectiveness and safety of thalidomide for treatment of oral and esophageal aphthous ulcers (those unrelated to a known infection or malignancy) in patients with advanced HIV disease. To evaluate the effect of thalidomide on HIV load in this patient population. Per 06/28/94 amendment, to evaluate the effectiveness of thalidomide in preventing recurrences in patients whose aphthae completely heal at the end of acute treatment.

SECONDARY: To evaluate the effect of thalidomide on blood tumor necrosis factor (TNF) levels and to obtain pharmacokinetic data on the drug. Per 06/28/94 amendment, to evaluate the safety of thalidomide. Per 05/10/95 amendment, to explore in a substudy the effects of thalidomide on idiopathic genital aphthous ulcers in HIV-infected women.

Aphthous ulcers of the mouth or esophagus can interfere with eating, resulting in malnutrition and wasting. Thalidomide has been proposed as an effective therapy for severe forms of aphthous ulceration in AIDS patients.

DETAILED DESCRIPTION:
Aphthous ulcers of the mouth or esophagus can interfere with eating, resulting in malnutrition and wasting. Thalidomide has been proposed as an effective therapy for severe forms of aphthous ulceration in AIDS patients.

Patients are randomized to receive 4 weeks of either thalidomide or placebo orally, administered once daily. Patients are followed weekly. Complete responders after 4 weeks of acute treatment enter a 24-week maintenance phase. A pharmacokinetic substudy will be included.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Anti-HIV therapy provided therapy has remained constant in the 4 weeks prior to study entry.
* Narcotic analgesia after the first week of treatment ONLY IF the patient is not experiencing somnolence.

Patients must have:

* Documented HIV infection or AIDS.
* Biopsy-confirmed aphthous ulceration of the mouth or esophagus lasting at least 2 weeks.
* Negative culture of ulcer for Herpes simplex.
* En face diameter of >= 5 mm for largest aphthous ulcer.
* Life expectancy of at least 3 months.

NOTE:

* This study is approved for prisoner participation.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known allergy to thalidomide.
* Grade 2 or worse bilateral peripheral neuropathy.

EXCLUDED FOR MAINTENANCE PHASE:

* Toxicity other than somnolence in acute phase that required discontinuation of drug.

Concurrent Medication:

Excluded:

* Acute therapy for opportunistic infection.
* ddC.
* Pentoxifylline.
* Methotrexate, trimetrexate, antineoplastic alkylating agents.
* Other putative immunomodulators.
* CNS depressants and/or medications with sedative or hypnotic effect.
* Systemic and/or oral topical corticosteroids.
* Systemic chemotherapy for Kaposi's sarcoma or other malignancies.
* Compounded antibacterial mouthwashes containing anti-infective agents (such as doxycycline, minocycline, tetracycline, or nystatin).

Concurrent Treatment:

Excluded:

* Radiation to head and/or neck.

Patients with the following prior conditions are excluded:

* History of grade 2 or worse bilateral peripheral neuropathy.
* Change in anti-HIV therapy within 4 weeks prior to study entry.
* Prior enrollment in ACTG 251 or prior treatment of aphthous ulcers with thalidomide.

Prior Medication:

Excluded:

* Systemic and/or oral topical corticosteroids within 1 week prior to first set of bloods drawn.
* Other putative immunomodulators within 2 weeks prior to study entry.
* Prior thalidomide for aphthous ulcers.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 164
Dates: Study Completion 1998-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobson JM, Study Chair
Locations (40):
- United States (39):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Illinois Masonic Med Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Comprehensive Health Care Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Adolescent AIDS Prog / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Drug Treatment Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Family Health Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - North Central Bronx Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Meharry Med College, Nashville, Tennessee
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Jacobson JM, Spritzler J, Fox L, Fahey JL, Jackson JB, Chernoff M, Wohl DA, Wu AW, Hooton TM, Sha BE, Shikuma CM, MacPhail LA, Simpson DM, Trapnell CB, Basgoz N. Thalidomide for the treatment of esophageal aphthous ulcers in patients with human immunodeficiency virus infection. National Institute of Allergy and Infectious Disease AIDS Clinical Trials Group. J Infect Dis. 1999 Jul;180(1):61-7. doi: 10.1086/314834. PMID 10353862
- [Background] Jacobson JM, Greenspan JS, Spritzler J, Ketter N, Fahey JL, Jackson JB, Fox L, Chernoff M, Wu AW, MacPhail LA, Vasquez GJ, Wohl DA. Thalidomide for the treatment of oral aphthous ulcers in patients with human immunodeficiency virus infection. National Institute of Allergy and Infectious Diseases AIDS Clinical Trials Group. N Engl J Med. 1997 May 22;336(21):1487-93. doi: 10.1056/NEJM199705223362103. PMID 9154767
- [Background] Gilden D. Thalidomide and aphthous ulcers. GMHC Treat Issues. 1995 Nov;9(11):12. PMID 11362988
- [Background] Jacobson JM, Greenspan JS, Spritzler J, Fox L, Fahey JL, Jackson JB, Chernoff M, Wohl DA, Pulvirenti JJ, Hooton TM, Shikuma C. Thalidomide in low intermittent doses does not prevent recurrence of human immunodeficiency virus-associated aphthous ulcers. J Infect Dis. 2001 Jan 15;183(2):343-346. doi: 10.1086/317928. Epub 2000 Dec 15. PMID 11120935
- [Background] Aweeka F, Trapnell C, Chernoff M, Jayewardene A, Spritzler J, Bellibas SE, Lizak P, Jacobson J. Pharmacokinetics and pharmacodynamics of thalidomide in HIV patients treated for oral aphthous ulcers: ACTG protocol 251. AIDS Clinical Trials Group. J Clin Pharmacol. 2001 Oct;41(10):1091-7. doi: 10.1177/00912700122012698. PMID 11583477